CLINICAL TRIAL: NCT01186445
Title: Evaluation of the Cardioprotective Effect of Intracoronary Injection of Morphine During Reperfusion in Acute Myocardial Infarction
Brief Title: Morphine In Acute Myocardial Infarction
Acronym: MIAMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIAMI-2008-09
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Cardioprotective effect; Pharmacological postconditioning; Morphine Chlorhydrate; Cardiac MRI
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine chlorhydrate (Experimental): Intracoronary injection of morphine chlorhydrate during reperfusion
  Interventions: Drug: morphine chlorhydrate
- Saline solution (Placebo Comparator): Intracoronary injection of saline solution during reperfusion
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: morphine chlorhydrate — 1mg of morphine chlorhydrate dilute in 3ml of saline solution, intracoronary injection, just before reperfusion
  Other Names: Morphine Chlorhydrate Lavoisier
  Arms: Morphine chlorhydrate
Drug: saline solution — 3 ml of saline solution , intracoronary injection during reperfusion
  Arms: Saline solution

SUMMARY:
The purpose of this study is to determine whether intracoronary injection of morphine chlorhydrate is effective to limit ischemia-reperfusion lesion during percutaneous coronary angioplasty in patients with acute myocardial infarction (AMI).

ELIGIBILITY:
Inclusion Criteria:

1. Acute Myocardial Infarction less than 6 hours defined by

   1. prolonged chest pain (>15 min)
   2. in association with

      * ST elevation 1mm or more in two contiguous leads
      * or occurence of Q wave in three contiguous leads
      * or occurence of left bundle branch block
2. Culprit lesion eligible for percutaneous coronary intervention (PCI)
3. TIMI flow 0 before PCI

Exclusion Criteria:

1. Fibrinolysis
2. Allergy to morphine
3. Active epilepsy
4. Brain injury or intracranial hypertension
5. Previous AMI, coronary artery bypass graft (CABG)
6. Cardiac arrest
7. Cardiogenic shock, significant mitral regurgitation or intraventricular communication at inclusion
8. Mechanical ventilation at inclusion
9. Significant ventricular arrhythmia or atrioventricular block type II or III at inclusion
10. Decompensated chronic obstructive pulmonary disease at inclusion
11. chronic hepatocellular failure
12. MRI contraindications
13. Gadolinium chelates injection contraindications
14. Current treatment with morphine chlorhydrate, buprenorphine, nalbuphine, pentazocine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Infarct size evaluated by delayed enhancement-magnetic resonance imaging | between day 3 and day 5 after acute myocardial infarction (AMI)

SECONDARY OUTCOMES:
Infarct size/area at risk ratio evaluated by MRI | between day 3 and day 5 after AMI
release of creatine kinase (CK) and troponin I (TnI) during reperfusion | during the first 72 hours after reperfusion
  The Area Under the Curve of CK and TnI during reperfusion
the Thrombolysis In Myocardial Infarction (TIMI) myocardial Blush after reperfusion | at day 0
ST segment resolution after reperfusion | during the first 24 hours after reperfusion
Left Ventricular Ejection Fraction measured by echocardiography | at day 1 and day 6
Infarct size measurement by delayed enhancement-magnetic resonance imaging | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lecorvoisier, MD, Principal Investigator — Henri Mondor University Hospital
Locations (2):
- France (2):
  - Henri Mondor Hospital, Créteil
  - Hopital Marie Lannelongue, Le Plessis-Robinson

REFERENCES:
- [Derived] Le Corvoisier P, Gallet R, Lesault PF, Audureau E, Paul M, Ternacle J, Ghostine S, Champagne S, Arrouasse R, Bitari D, Mouillet G, Dubois-Rande JL, Berdeaux A, Ghaleh B, Deux JF, Teiger E. Intra-coronary morphine versus placebo in the treatment of acute ST-segment elevation myocardial infarction: the MIAMI randomized controlled trial. BMC Cardiovasc Disord. 2018 Oct 19;18(1):193. doi: 10.1186/s12872-018-0936-8. PMID 30340532